CLINICAL TRIAL: NCT03198559
Title: Combination Latency Reversal With High Dose Disulfiram Plus Vorinostat in HIV-infected Individuals on ART (DIVA): A Single Arm Clinical Trial
Brief Title: Combination Latency Reversal With High Dose Disulfiram Plus Vorinostat in HIV-infected Individuals on ART
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: A re-evaluation of research risks to participants were greater than originally anticipated
Sponsor: University of Melbourne (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); The Alfred (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSD IIS-55750
Record Dates: First submitted 2017-06-14; First posted 2017-06-26 (Actual); Results first posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2023-06

CONDITIONS: HIV Infections
Keywords: HIV latency; Disulfiram; Vorinostat; Latency Reversing Agents; Histone Deacetylase Inhibitors (HDACi)
MeSH Terms: conditions — HIV Infections | interventions — Disulfiram; Vorinostat

STUDY DESIGN:
Intervention Model Description: Single arm, single site,
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Participants current ART regimen:
  2 grams disulfiram by mouth per day for a total of 28 days
  400mg vorinostat by mouth per day on days 8, 9,10 and days 22, 23, 24
  Interventions: Drug: Disulfiram, (National Drug Code) NDC 0378-4141-01; Drug: Vorinostat, NDC 00006-0568-40

INTERVENTIONS:
Drug: Disulfiram, (National Drug Code) NDC 0378-4141-01 — This study will provide open label disulfiram. Participants will take 2 grams (4x500mg tablets) of disulfiram per day for a total of 28 days
Drug: Vorinostat, NDC 00006-0568-40 — This study will provide open label vorinostat. Participants will take 400mg (4x100mg capsules) of vorinostat per day on days 8, 9, 10 and days 22, 23, 24.
  Other Names: Zolinza

SUMMARY:
Antiretroviral therapy (ART) dramatically reduces Human Immunodeficiency Virus (HIV) replication leading to restoration of immune function and a near normal life expectancy, but treatment is lifelong and there is no cure. The major barrier to a cure is the persistence of long lived cluster of differentiation 4 (CD4+) T-cells that contain a "silenced" form of HIV, called HIV latency.

The purpose of this research is to investigate whether it may be possible to reduce the amount of dormant HIV infection in immune cells, by "turning on" or activating the virus and hence force it out of the latently infected memory T cells. This leads to production of HIV by the cell, which will either die or will be recognized and eliminated by the immune system. As very few T cells are latently infected with HIV, the death of these cells is not expected to affect the function of the immune system and further infection of new cells is expected to be prevented by ART.

DETAILED DESCRIPTION:
One strategy aimed at reducing the frequency of latently infected cells in HIV-infected individuals on antiretroviral therapy (ART) is the use of pharmacological agents to reverse HIV latency, thereby initiating virus-mediated cell lysis or immune-mediated killing. Recent clinical trials of latency reversing agents (LRAs) in HIV infected subjects on ART, including histone deacetylase inhibitors (HDACi) and the anti-alcoholism drug disulfiram, have shown that inducing an increase in Cell Associated Unspliced (CA-US) HIV RNA or plasma HIV RNA is possible. Yet, these interventions did not have a demonstrable effect on the frequency of latently infected cells or time to viral rebound after cessation of ART, potentially because latency reversal alone didn't trigger an adequate immune response or cell death or that the potency of latency reversal with a single-agent intervention over a very short period of time, lacked sufficient potency, as suggested by recent in vitro studies. It is highly likely that long-term remission off ART will require interventions that lead to both a reduction in latently infected cells and an increase in HIV-specific immunity, therefore identifying a strategy to increase viral antigens on the surface of latently infected cells will be a key component of this strategy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years with documented HIV-1 infection (antibody positive or detectable plasma HIV-1 RNA)
* Receiving combination ART with plasma HIV RNA <50 copies/mL for >3 years
* CD4+ T cell count >350 microliter at screening
* Able to provide informed consent
* Willing to abstain from alcohol consumption from one day before to 14 days after completing 28 days of disulfiram
* One month post influenza vaccine (from screening visit)
* Women of non-child-bearing potential defined as > 12 months of spontaneous amenorrhea and ≥ 45 years of age, or documented medical history of one of the following: hysterectomy, bilateral oophorectomy or tubal ligation.
* Women of Child Bearing Potential (WOCBP) with a negative pregnancy test at Screening and agrees to use one of the study protocol specified methods of contraception to avoid pregnancy

Exclusion Criteria:

* Current alcohol use disorder or hazardous alcohol use (>7 drinks per week for women or > 14 drinks per week for men) as determined by clinical evaluation
* Current or recent (in the last 4 days) use of metronidazole or any drug formulation that contains alcohol or that might contain alcohol, including the gelatin capsule and liquid formulations of ritonavir, ritonavir/lopinavir, amprenavir and fosamprenavir, and alcohol-containing preparations such as cough syrups, tonics etc.
* Current use of tipranavir or Maraviroc
* Current use of zidovudine, stavudine or didanosine (as disulfiram potentially has potent irreversible inhibitory effects on mitochondrial metabolism and hence could exacerbate the toxicity of these drugs)
* Concurrent use of rivaroxaban (a CYP3A metabolized medication) as the cytochrome P450 inhibitory effects of disulfiram on rivaroxaban are unknown
* Current use of warfarin
* Individuals who intend to modify antiretroviral therapy during the study period for any reason
* Significant myocardial disease (current myocarditis or reduced left ventricular ejection fraction below the lower limit of normal) or diagnosed coronary artery disease
* Significant renal disease (eGFR <50 milliliter/minute)
* History of psychosis, seizure disorder, abnormal electroencephalogram or brain damage with significant persisting neurological deficit
* Prior malignancy active within the previous 3 years except for local curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the prostate, cervix or breast.
* Known hypersensitivity to disulfiram or vorinostat or contraindications to treatment with these agents
* Participation in another latency reversal study or receipt of vorinostat or disulfiram in the previous 12 months before starting the investigational treatment
* Any significant acute medical illness requiring hospitalization within preceding 8 weeks
* Hepatitis B (HBV) or hepatitis C (HCV) co-infection as determined by detection of HBsAg or HCV RNA (Individuals with prior hepatitis infection that is now cleared are eligible for enrolment)
* Receipt of immunomodulating agents (excluding immunization) or systemic chemotherapeutic agents within 28 days prior to study entry
* Current or recent gastrointestinal disease or surgery that may impact the absorption of the investigational drug
* Active substance use that in the opinion of the investigator will prevent adequate compliance with study procedures
* Women who are currently pregnant or breastfeeding
* Women of Child Bearing Potential (WOCBP) who are unwilling or unable to use an acceptable method of contraception to avoid pregnancy
* Unable or unwilling to adhere to protocol procedures
* The following laboratory values within 6 weeks before starting the investigational drug (lab tests may be repeated to obtain acceptable values before failure at screening is concluded)

  * Hepatic transaminases (AST or ALT) ≥3 x upper limit of normal (ULN)
  * Serum total bilirubin ≥1.5 x ULN
  * eGFR <50 milliliter/min
  * Hemoglobin <11.0 g/deciliter
  * Platelet count ≤100 x10^9/L (liter)
  * Absolute neutrophil count ≤1.5x10^9/L
  * Serum potassium, magnesium, phosphorus outside normal limits
  * Total calcium (corrected for serum albumin) or ionized calcium ≤ lower normal limits

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2019-04-09 (Actual); Study Completion 2019-04-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon R Lewin, FRACP, PhD, Principal Investigator — The Doherty Institute, University of Melbourne
Locations (1):
- Department of Infectious Diseases, Alfred Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data

REFERENCES:
- [Result] McMahon JH, Evans VA, Lau JSY, Symons J, Zerbato JM, Chang J, Solomon A, Tennakoon S, Dantanarayana A, Hagenauer M, Lee S, Palmer S, Fisher K, Bumpus N, Heck CJS, Burger D, Wu G, Zuck P, Howell BJ, Zetterberg HH, Blennow K, Gisslen M, Rasmussen TA, Lewin SR. Neurotoxicity with high-dose disulfiram and vorinostat used for HIV latency reversal. AIDS. 2022 Jan 1;36(1):75-82. doi: 10.1097/QAD.0000000000003091. PMID 34586085

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment began August 8, 2017. Participants were enrolled for screening between this date and when recruitment into the study was suspended on October 19, 2017. In the end, 5 participants were consented into the study and found eligible to begin treatment. Only 2 participants received treatment before the study was suspended.
Pre-assignment Details: Enrolled participants who were screened and found eligible to begin on-study treatment were started in a staggered-start. Essentially this meant that the first 2 eligible participants started treatment at the same time. Only once the treatment phase had been completed would the next 2 eligible participants begin the on-study treatment phase.
Groups:
- Treatment: Participants would receive
  2 grams disulfiram by mouth per day for a total of 28 days
  400mg vorinostat by mouth per day on days 8, 9,10 and days 22, 23, 24
  Disulfiram, (National Drug Code) NDC 0378-4141-01: This study will provide open label disulfiram. Participants will take 2 grams (4x500mg tablets) of disulfiram per day for a total of 28 days
  Vorinostat, NDC 00006-0568-40: This study will provide open label vorinostat. Participants will take 400mg (4x100mg capsules) of vorinostat per day on days 8, 9, 10 and days 22, 23, 24.
Period: Overall Study
Arm/Group | Treatment
Started | 2
Completed | 0
Not Completed | 2
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Groups:
- Experimental: Participants current ART regimen:
  2 grams disulfiram by mouth per day for a total of 28 days
  400mg vorinostat by mouth per day on days 8, 9,10 and days 22, 23, 24
  Disulfiram, (National Drug Code) NDC 0378-4141-01: This study will provide open label disulfiram. Participants will take 2 grams (4x500mg tablets) of disulfiram per day for a total of 28 days
  Vorinostat, NDC 00006-0568-40: This study will provide open label vorinostat. Participants will take 400mg (4x100mg capsules) of vorinostat per day on days 8, 9, 10 and days 22, 23, 24.
Arm/Group | Experimental
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Australia | 2

OUTCOME MEASURES:

1. Primary Outcome: Day 11 Plasma HIV RNA Relative to Baseline
Description: The primary endpoint was to determine the change from baseline to day 11 of plasma HIV RNA levels after 11 continuous days of disulfiram with administration of vorinostat on days 8, 9 and 10 in HIV infected individuals on suppressive ART.
Time Frame: Baseline and 11 days
Population: The analysis included all participants who received at least one dose of study drug.
Measure: Number; unit: Fold change from baseline to day 11
Arm/Group | Experimental
Number analyzed (Participants) | 2
Fold change from baseline to day 11
  Participant 1: number analyzed (Participants) | 1
  Participant 1 | 1
  Participant 2: number analyzed (Participants) | 1
  Participant 2 | 13.5

2. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events
Description: This secondary outcome was to determine the Incidence of treatment-emergent adverse events [Safety and Tolerability] during a 28 day course of continuous disulfiram with intermittent administration of 3 days of vorinostat on two occasions in HIV infected individuals on suppressive ART.
  An adverse event is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that; results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations as judged by physician.
  Systematic assessments of adverse events were performed at each visit, including unscheduled visits
Time Frame: Adverse events were collected continuously throughout the study duration from day 1 on treatment until 2 months since last dose of study drug, an average duration of 3 months
Population: All participants who received one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 2
Participants
  Any SAE | 2
  Any non-SAE | 2

3. Secondary Outcome: Plasma HIV RNA Relative to Baseline at Additional Time Points
Description: This secondary outcome was to determine the fold change in plasma HIV RNA levels at additional time points during and after 11 continuous days of disulfiram with administration of vorinostat on days 8, 9 and 10 in HIV infected individuals on suppressive ART.
Time Frame: Baseline to Days 8, 15, 21, 38, 59, 196, 197. Data is reported for days where samples were collected for each participant.
Population: All participants who received at least one dose of treatment was analyzed.
Measure: Number; unit: Fold change from baseline
Arm/Group | Experimental
Number analyzed (Participants) | 2
Fold change from baseline
  Participant 1 - Day 8: number analyzed (Participants) | 1
  Participant 1 - Day 8 | 1
  Participant 1 - Day 59: number analyzed (Participants) | 1
  Participant 1 - Day 59 | 1
  Participant 1 - Day 197: number analyzed (Participants) | 1
  Participant 1 - Day 197 | 1
  Participant 2 - Day 8: number analyzed (Participants) | 1
  Participant 2 - Day 8 | 9.9
  Participant 2 - Day 15: number analyzed (Participants) | 1
  Participant 2 - Day 15 | 14.4
  Participant 2 - Day 21: number analyzed (Participants) | 1
  Participant 2 - Day 21 | 45.9
  Participant 2 - Day 38: number analyzed (Participants) | 1
  Participant 2 - Day 38 | 18.3
  Participant 2 - Day 196: number analyzed (Participants) | 1
  Participant 2 - Day 196 | 5

4. Other Pre Specified Outcome: HIV RNA Transcription Relative to Baseline at Additional Time Points
Description: This secondary outcome was to measure HIV transcription measured by cell-associated unspliced HIV RNA (CA-US HIV RNA) in peripheral blood CD4+ T cells relative to baseline
Time Frame: Baseline to Days 8, 11, 15, 21, 38, 59, 196, 197. Data is reported for days where samples were collected for each participant.
Population: All participants who had received at least 1 dose of treatment
Measure: Number; unit: Fold change from baseline
Arm/Group | Experimental
Number analyzed (Participants) | 2
Fold change from baseline
  Participant 1 - Day 8: number analyzed (Participants) | 1
  Participant 1 - Day 8 | 3.33
  Participant 1 - Day 11: number analyzed (Participants) | 1
  Participant 1 - Day 11 | 5.13
  Participant 1 - Day 59: number analyzed (Participants) | 1
  Participant 1 - Day 59 | 4.56
  Participant 1 - Day 197: number analyzed (Participants) | 1
  Participant 1 - Day 197 | 12.72
  Participant 2 - Day 8: number analyzed (Participants) | 1
  Participant 2 - Day 8 | 1.56
  Participant 2 - Day 11: number analyzed (Participants) | 1
  Participant 2 - Day 11 | 0.91
  Participant 2 - Day 15: number analyzed (Participants) | 1
  Participant 2 - Day 15 | 0.64
  Participant 2 - Day 21: number analyzed (Participants) | 1
  Participant 2 - Day 21 | 0.72
  Participant 2 - Day 38: number analyzed (Participants) | 1
  Participant 2 - Day 38 | 0.41
  Participant 2 - Day 196: number analyzed (Participants) | 1
  Participant 2 - Day 196 | 3.77

5. Other Pre Specified Outcome: Cell Associated Total HIV DNA Relative to Baseline at Additional Points
Description: This outcome was to measure Cell-associated total and integrated HIV DNA in peripheral blood CD4+ T cells relative to baseline
Time Frame: Baseline and Days 38, 59, 196 and 197. Data is reported for days where results are available for each participant.
Population: All participants who received at least one dose of treatment
Measure: Number; unit: Fold change from baseline
Arm/Group | Treatment
Number analyzed (Participants) | 2
Fold change from baseline
  Participant 1 - Day 59: number analyzed (Participants) | 1
  Participant 1 - Day 59 | 0.7
  Participant 1 - Day 197: number analyzed (Participants) | 1
  Participant 1 - Day 197 | 0.72
  Participant 2 - Day 38: number analyzed (Participants) | 1
  Participant 2 - Day 38 | 0.74
  Participant 2 - Day 196: number analyzed (Participants) | 1
  Participant 2 - Day 196 | 1.72

6. Other Pre Specified Outcome: Cell-associated Integrated HIV DNA Relative to Baseline at Additional Points
Description: This outcome was to measure cell-associated integrated HIV DNA in peripheral blood CD4+ T cells relative to baseline
Time Frame: Baseline to Days 38, 59, 197, 196. Data is reported for days where samples were collected for each participant.
Population: All participants who received at least one dose of treatment
Measure: Number; unit: Fold change from baseline
Arm/Group | Treatment
Number analyzed (Participants) | 2
Fold change from baseline
  Participant 1 - Day 59: number analyzed (Participants) | 1
  Participant 1 - Day 59 | 1.47
  Participant 1 - Day 197: number analyzed (Participants) | 1
  Participant 1 - Day 197 | 2.52
  Participant 2 - Day 38: number analyzed (Participants) | 1
  Participant 2 - Day 38 | 0.37
  Participant 2 -Day 196: number analyzed (Participants) | 1
  Participant 2 -Day 196 | 1.46

7. Other Pre Specified Outcome: HIV Levels Relative to Baseline
Description: This outcome was to measure the frequency of inducible virus as measured by Tat/rev limiting dilution assay (TILDA) in peripheral blood CD4+ T cells relative to baseline.
  Not conducted as part of the analysis and there are no future plans to assess this outcome, as analysis from 2 participants would not provide any meaningful results, given that the participants did not manage to complete the treatment course.
Time Frame: Day 56
Population: This primary endpoint was not performed. See outcome measure description for reasoning
Arm/Group | Treatment
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Vorinostat Concentration in Plasma
Description: This outcome was to measure the concentrations of vorinostat (including its metabolites) in plasma.
Time Frame: Baseline and days 8, 11, 15, 21, 37, 58. Data is reported for days where samples were collected for each participant.
Population: All participants who received at least one dose of treatment.
Measure: Number; unit: ng/mL
Arm/Group | Experimental
Number analyzed (Participants) | 2
ng/mL
  Participant 1 - Baseline: number analyzed (Participants) | 1
  Participant 1 - Baseline | NA — Concentration was below limit of detection for assay (<2.00 ng/mL)
  Participant 1 - Day 8: number analyzed (Participants) | 1
  Participant 1 - Day 8 | NA — Concentration was below limit of detection for assay (<2.00 ng/mL)
  Participant 1 - Day 11 | 6.52
  Participant - Day 58 | NA — Concentration was below limit of detection for assay (<2.00 ng/mL)
  Participant 2 - Baseline | NA — Concentration was below limit of detection for assay (<2.00 ng/mL)
  Participant 2 - Day 8 | NA — Concentration was below limit of detection for assay (<2.00 ng/mL)
  Participant 2 - Day 11 | 7.6
  Participant 2 - Day 15 | NA — Concentration was below limit of detection for assay (<2.00 ng/mL)
  Participant 2 - Day 21 | NA — Concentration was below limit of detection for assay (<2.00 ng/mL)
  Participant 2 - Day 38 | NA — Concentration was below limit of detection for assay (<2.00 ng/mL)

9. Other Pre Specified Outcome: Disulfiram Concentration in Plasma
Description: This outcome was to measure the concentrations of disulfiram (including its metabolites) in plasma
Time Frame: Days 8, 11, 22, 25, 28, 56 and 196 Data is reported for days where samples were collected for each participant.
Population: All participants who received at least one dose of treatment.
Measure: Number; unit: ng/mL
Arm/Group | Experimental
Number analyzed (Participants) | 2
ng/mL
  Participants 1 and 2 - Day 8 | NA — Concentration below limit of detection
  Participants 1 and 2 - Day 11 | NA — Concentration below limit of detection
  Participant 1 - Day 58: number analyzed (Participants) | 1
  Participant 1 - Day 58 | NA — Concentration below limit of detection
  Participant 2 -Day 15: number analyzed (Participants) | 1
  Participant 2 -Day 15 | NA — Concentration below limit of detection
  Participant 2 - Day 21: number analyzed (Participants) | 1
  Participant 2 - Day 21 | NA — Concentration below limit of detection

10. Other Pre Specified Outcome: p24 Expression in CD4+ T-cells Relative to Baseline
Description: This outcome was to measure the p24 expression in CD4+ T-cells relative to baseline
Time Frame: Baseline and Days 8, 11, 15, 21, 37, 58, 196 and 197. Data is reported for days where samples were collected for each participant.
Population: All participants who received at least one dose of treatment.
Measure: Number; unit: Fold change from baseline
Arm/Group | Treatment
Number analyzed (Participants) | 2
Fold change from baseline
  Participant 1 - Day 8: number analyzed (Participants) | 1
  Participant 1 - Day 8 | 0.83
  Participant 1 - Day 11 | 0.78
  Participant 1 - Day 58 | 2.13
  Participant 1 - Day 197 | 0.96
  Participant 2 - Day 8: number analyzed (Participants) | 1
  Participant 2 - Day 8 | 1.96
  Participant 2 - Day 11 | 0.91
  Participant 2 - Day 15 | 1.26
  Participant 2 - Day 21 | 1
  Participant 2 - Day 38 | 1.09
  Participant 2 - Day 196 | 1.39

ADVERSE EVENTS:
Time Frame: Adverse event data measured from Day 1 on treatment until two months post last day on treatment, for an average duration of 3 months.
Description: All Serious Adverse Events, and Other Adverse Events (non-serious) have been reported.
  Any abnormality was graded according to Division of Acquired Immunodeficiency Syndrome (DAIDS) toxicity scales from Grade 1 to 4 (1=Mild, 2=Moderate, 3=Severe, 4=Potentially life threatening) where known has been added
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 2/2
Serious Adverse Events (participants affected / at risk) | 2/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=2)
Altered mental status, Grade 3 (Nervous system disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=2)
Lethargy, all grades (Nervous system disorders) | 2
Alanine aminotransferase elevated, Grade 1 (Investigations) | 2
Diarrhea, grade 1 (Gastrointestinal disorders) | 1
Hematuria, grade 1 (Investigations) | 1
Dysgeusia, grade 1 (Nervous system disorders) | 1
Flu like symptoms, grade 2 (General disorders) | 1
thrombosis or embolism, grade 2 (Cardiac disorders) | 1
Fatigue, all grades (General disorders) | 2

LIMITATIONS AND CAVEATS:
Early termination of the study lead to a small numbers of participants analyzed. Therefore there was insufficient power to measure the effect of the intervention.

Other key limitations to this study include:

* only 2 participants received study drug;
* participants did not complete the full course of treatment as outlined in the study design;
* 1 participant missed Day 10 study medication, stopped study treatment on Day 17;
* 1 participant ceased study medication on Day 11;

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT03198559/Prot_SAP_000.pdf